CLINICAL TRIAL: NCT00301938
Title: A Phase 1 Study of UCN-01 in Combination With Perifosine in Patients With Relapsed and Refractory Acute Leukemias and High Risk MDS
Brief Title: 7-Hydroxystaurosporine and Perifosine in Treating Patients With Relapsed or Refractory Acute Leukemia, Chronic Myelogenous Leukemia or High Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00149; NCI-2009-00149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSGCC-0507; NCI-7311; MSGCC-H-27229-0507; CDR0000465368; GCC 0507 (Other: University of Maryland Greenebaum Cancer Center); 7311 (Other: CTEP)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Acute Promyelocytic Leukemia (M3); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Blastic Phase Chronic Myelogenous Leukemia; Myelodysplastic/Myeloproliferative Neoplasms; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; T-cell Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — 7-hydroxystaurosporine; perifosine; octadecyl-(N,N-dimethylpiperidino-4-yl)-phosphate

ARMS (2):
- Arm I (enzyme inhibitor, chemotherapy) (Experimental): Patients receive a loading dose of oral perifosine every 6 hours on day 1 followed by a maintenance dose once daily on days 2-28 of course 1 and then once daily on days 1-28 in all subsequent courses. Patients also receive 7-hydroxystaurosporine IV over 3 hours on day 4. Cohorts of 3-6 patients receive escalating doses of 7-hydroxystaurosporine until the MTD is determined.
  Interventions: Drug: 7-hydroxystaurosporine; Drug: perifosine; Other: pharmacological study
- Arm 2 (enzyme inhibitor, chemotherapy) (Experimental): Patients receive 7-hydroxystaurosporine IV over 3 hours on day 1 at the MTD determined in group I. Patients also receive oral perifosine as a loading dose every 6 hours on day 4 followed by a maintenance dose once daily on days 5-28 of course 1 and then once daily on days 1-28 in all subsequent courses.
  Interventions: Drug: 7-hydroxystaurosporine; Drug: perifosine; Other: pharmacological study

INTERVENTIONS:
Drug: 7-hydroxystaurosporine — Given IV
  Other Names: UCN-01
Drug: perifosine — Given orally
  Other Names: D21266; octadecylphosphopiperidine
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of 7-hydroxystaurosporine when given together with perifosine in treating patients with relapsed or refractory acute leukemia, chronic myelogenous leukemia, or myelodysplastic syndromes. 7-Hydroxystaurosporine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as perifosine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving 7-hydroxystaurosporine together with perifosine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define the maximum tolerated dose and recommended phase II dose of UCN-01 (7-hydroxystaurosporine) administered after perifosine in patients with relapsed or refractory acute leukemia, chronic myelogenous leukemia, or high risk myelodysplastic disorders.

SECONDARY OBJECTIVES:

I. Evaluate the safety and toxicity of UCN-01 administered after perifosine in these patients.

II. Evaluate the safety and toxicity of perifosine administered after UCN-01 in these patients.

III. Document responses in patients treated with this regimen. IV. Observe the pharmacokinetics of both perifosine and UCN-01 when administered in combination.

V. Study the pharmacodynamics of perifosine alone, UCN-01 alone, and in combination in leukemic blast cells.

OUTLINE: This is a multicenter, dose-escalation study of 7-hydroxystaurosporine. The first patients enrolled in the study are assigned to arm 1. Once the maximum tolerated dose (MTD) is determined in arm 1, subsequent patients are enrolled in arm 2.

ARM 1: Patients receive a loading dose of oral perifosine every 6 hours on day 1 followed by a maintenance dose once daily on days 2-28 of course 1 and then once daily on days 1-28 in all subsequent courses. Patients also receive 7-hydroxystaurosporine intravenously (IV) over 3 hours on day 4. Cohorts of 3-6 patients receive escalating doses of 7-hydroxystaurosporine until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

ARM 2: Patients receive 7-hydroxystaurosporine IV over 3 hours on day 1 at the MTD determined in group I. Patients also receive oral perifosine as a loading dose every 6 hours on day 4 followed by a maintenance dose once daily on days 5-28 of course 1 and then once daily on days 1-28 in all subsequent courses. In both groups, treatment repeats every 28 days for ≥ 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete remission (CR) or a CR with incomplete hematologic recovery receive 4 additional courses beyond documentation of CR. Patients who achieve a partial remission or hematologic improvement may continue treatment in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hematologic malignancy of 1 of the following types:

  * Relapsed or refractory acute myelogenous leukemia (AML)

    * Patients with acute promyelocytic leukemia t(15;17) are eligible provided they failed a prior tretinoin and arsenic-containing regimen

      * Patients should be either refractory to both agents (absence of durable hematologic response) OR relapsed after a complete response duration of < 6 months
  * Relapsed or refractory pre-B-cell or T-cell acute lymphoblastic leukemia (ALL)
  * Chronic myelogenous leukemia (CML) in accelerated or blastic phase that is refractory to imatinib mesylate

    * Must have evidence of disease progression despite continued treatment with imatinib mesylate
  * AML arising in the setting of underlying myelodysplastic syndromes (MDS) and/or myeloproliferative disorders (MPD)
  * Secondary or therapy-related AML
  * De novo AML or pre-B-cell or T-cell ALL in adults > 60 years of age with poor-risk features, such as complex (≥ 3) or adverse cytogenetics

    * The following are considered adverse cytogenetic abnormalities for AML:

      * -5q
      * 7q-
      * 9q-
      * 20q-
      * abn12p
      * +21
      * +8
      * t(6;9)
      * t(6;11)
      * t(11;19)
      * -7
      * -5
      * inv3/t(3;3)
      * abn11q23
      * abn17p
      * abn21q
      * t(9;22) refractory to imatinib mesylate
    * The following are considered adverse cytogenetic abnormalities for ALL:

      * t(9;22) refractory to imatinib mesylate
      * Hypodiploidy
      * t(4;11)
      * t(1;19)
  * Myelodysplastic Syndromes (MDS) meeting 1 of the following criteria:

    * Intermediate and high risk (i.e., International Prognostic Scoring System [IPSS] ≥ 1.5) MDS that is refractory or has progressed after treatment with azacitidine and/or decitabine
    * Intermediate and high risk (i.e., IPSS ≥ 1.5) MDS with a 5q- cytogenetic abnormality that is refractory or has progressed after treatment with lenalidomide, azacitidine, or decitabine
    * Intermediate 2 and high risk MDS without 5q- cytogenetic abnormality that is refractory or has progressed after azacitidine or decitabine

      * Original 5q must also be refractory to lenalidomide
* Received OR ineligible for established curative regimens, including stem cell transplantation
* No active CNS leukemia
* ECOG performance status (PS) 0-2 OR Karnofsky PS ≥ 60%
* Total or direct bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN
* Creatinine ≤ 2 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No hyperleukocytosis (i.e., WBC > 30,000/mm^3) (recent treatment with hydroxyurea to prevent impending leukostasis allowed provided there has been no dose increase for ≥ 1 week)
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to UCN-01 or perifosine
* No intrinsic impaired organ function
* No active, uncontrolled infection

  * Infection that is controlled with antibiotics allowed
* No symptomatic cardiac disease
* No active ischemia on EKG
* LVEF ≥ 40% by echocardiogram or MUGA

  * Patients with a history of cardiac disease or mediastinal radiation should undergo testing of ventricular function
* No poorly controlled diabetes mellitus
* No psychiatric illness or social situation that would preclude giving informed consent or complying with study requirements
* No HIV positivity
* See Disease Characteristics
* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for carmustine or mitomycin C) and recovered
* At least 4 weeks since prior radiotherapy and recovered
* At least 4 weeks since prior autologous stem cell transplantation (SCT)
* At least 90 days since prior allogeneic SCT

  * No evidence of graft vs host disease
* At least 2 weeks since prior immunosuppressive therapy
* No concurrent hematopoietic growth factors or biologic agents
* No other concurrent investigational agents, chemotherapy, radiotherapy, or immunotherapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-12; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of 7-hydroxystaurosporine administered after perifosine | Course 1 (first 28 days)
  Evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The highest dose with none or one DLT observed in six patients will be declared as MTD. To ensure the toxicity at the MTD is acceptable, additional 6 patients will be accrued at the MTD.

SECONDARY OUTCOMES:
Response rate, determined by improvement of blast cell count, degree of marrow infiltration by tumor cells, and improvement in peripheral blood count | Baseline, at the end of course 1 (day 21-28), and any time that disease progression is suspected
  For patients with acute leukemias we will use revised International Working Group (IWG) response criteria as published by Cheson et al. For patients with MDS we will use IWG response assessment for MDS. 90% confidence interval (CI) will be provided.
Progression free survival | The time between the study entry and the first date that relapse or progressive disease is objectively documented, or death from any cause occurs
  Estimated using the Kaplan-Meier method.
Disease specific survival and survival Rate | 1 year
  Estimated using the Kaplan-Meier method.
Overall survival | From time of enrollment onto this study to the time of death
  Estimated using the Kaplan-Meier method.
Pharmacokinetics and pharmacodynamics of both perifosine and 7-hydroxystaurosporine | Baseline and at weeks 1, 5, and 9
  Descriptive statistics and confidence intervals will be provided for molecular endpoints of drugs action: total akt, phospho akt, total erk, phospho erk, p21 in peripheral blood and marrow. We will also dichotomize pharmacokinetic levels at the median, and estimate differences in response rates for high versus low levels, using Fisher's exact test at the one-sided 0.05 significance level.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gojo, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Gojo I, Perl A, Luger S, Baer MR, Norsworthy KJ, Bauer KS, Tidwell M, Fleckinger S, Carroll M, Sausville EA. Phase I study of UCN-01 and perifosine in patients with relapsed and refractory acute leukemias and high-risk myelodysplastic syndrome. Invest New Drugs. 2013 Oct;31(5):1217-27. doi: 10.1007/s10637-013-9937-8. Epub 2013 Feb 27. PMID 23443507